CLINICAL TRIAL: NCT01043562
Title: Defibrillation Thresholds in a Pediatric Cohort Using Binary Search Protocol
Brief Title: Precise Measurement of Pediatric Defibrillation Thresholds
Status: Completed | Type: Observational
Sponsor: Boston Children's Hospital (Other)
Responsible Party: Principal Investigator, Andrew Eric Radbill, Assistant Professor of Pediatrics, Boston Children's Hospital
Other Study IDs: 09-04-0209
Record Dates: First submitted 2010-01-06; First posted 2010-01-07 (Estimated); Results first posted 2018-02-05 (Actual); Last update posted 2018-02-05 (Actual); Status verified 2017-07

CONDITIONS: Pediatrics; Defibrillators, Implantable

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Pediatric ICD pts: Inclusion criteria for study participants included: 1) weight ≤60 kg, 2) new or existing ICD system, and 3) clinically necessary assessment of the defibrillation efficacy of the ICD system. Transvenous systems utilized a high-voltage ICD coil with active-fixation lead attached to the right ventricular endocardial surface, whereas non-transvenous systems depended upon a high-voltage shocking coil placed within the pericardial, subcutaneous or pleural space. To be included in the post-shock pacing portion of the study, adequate sinus and AV node function had to be present at baseline. Exclusion criteria included 1) tenuous hemodynamic status felt to warrant abbreviation of the defibrillation efficacy testing or 2) inability to induce fibrillation during defibrillation threshold testing (DFT).
  Interventions: Diagnostic Test: Defibrillator threshold testing; Other: Observation of post-shock intrinsic cardiac rhythm

INTERVENTIONS:
Diagnostic Test: Defibrillator threshold testing — Measurement of the defibrillation threshold was performed using a modified binary search protocol. This protocol specified three distinct inductions of ventricular fibrillation (VF) for all subjects, with a 3-5 minute observation/waiting period between inductions. The initial shock energy was programmed at 9 joules (J) for all patients, with internal rescue shocks at 31J followed by device-specific maximum deliverable energy. The outcome of the initial induction determined the programmed energies for both the initial and internal rescue shocks for the second induction, and likewise for the third induction. All shocks were biphasic and delivered at manufacturers' default tilt, polarity and duration, and all final programmed shock vectors included an active can. External defibrillation pads were in place for delivery of external rescue shock should the internal shocks fail.
Other: Observation of post-shock intrinsic cardiac rhythm — Prior to each of the three ventricular fibrillation inductions performed as part of the binary search protocol, post-shock pacing was re-programmed using a pre-determined, stepwise protocol that progressively decreased the lower rate limit. For the purpose of this protocol, post-shock pacing was considered necessary if 1) ≥7 ventricular-paced beats or 2) asystole >4 seconds was observed in the first 20 seconds after defibrillation, or if the systolic blood pressure demonstrated a >10% decrease from pre-induction baseline at follow-up measurement 1 minute post-defibrillation. Rescue ventricular pacing via the programmer was available for all subjects.

SUMMARY:
Patients who receive an implantable cardioverter-defibrillator (ICD) usually undergo testing at the end of the ICD procedure to measure the amount of energy able to successfully defibrillate the heart (defibrillation threshold testing, or DFT). This study proposes to perform that measurement in pediatric patients already undergoing clinically necessary ICD procedures, with the measurement performed using a binary search method that has been previously validated in adult cohorts. We hypothesize that pediatric DFTs, when precisely measured, may be lower than previously assumed from extrapolation of adult data.

ELIGIBILITY:
Inclusion Criteria:

* Current follow-up at Children's Hospital Boston
* Children with current or planned ICDs who are scheduled by their primary electrophysiologist for clinically necessary assessment/re-assessment of defibrillation threshold
* If the patient has an ICD system with a non-transvenous shock coil: weight ≤35kg at time of initial implant, with current weight <50kg
* If the patient has an ICD system with a conventional transvenous shock coil: current weight ≤60kg

Exclusion Criteria:

* Clinical failure of any system component not able to be addressed by hardware repair or exchange
* Hemodynamic instability that in the judgment of the primary electrophysiologist warrants abbreviation of DFT assessment
* Unsuccessful induction of fibrillation during DFT testing

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: All patients seen by the electrophysiology service at Children's Hospital Boston who are identified to be at very high risk of sudden cardiac death and in need of an ICD
Sampling Method: Non-Probability Sample
Enrollment: 20 (Actual)
Dates: Start 2009-06-04 (Actual); Primary Completion 2010-05-26 (Actual); Study Completion 2012-05-10 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Andrew E Radbill, MD, Principal Investigator — Boston Children's Hospital
Locations (1):
- Children's Hospital Boston, Boston, Massachusetts, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Groups:
- Pediatric ICD Pts: Inclusion criteria: 1) weight ≤60 kg, 2) new or existing ICD system, and 3) clinically necessary assessment of the defibrillation efficacy of the ICD system. Transvenous systems utilized a high-voltage ICD coil with active-fixation lead attached to the right ventricular endocardial surface, whereas non-transvenous systems depended upon a high-voltage shocking coil placed within the pericardial, subcutaneous or pleural space. To be included in the post-shock pacing portion of the study, adequate sinus and AV node function had to be present at baseline. Exclusion criteria included 1) tenuous hemodynamic status felt to warrant abbreviation of the defibrillation efficacy testing or 2) inability to induce fibrillation during defibrillation threshold testing (DFT).
  Defibrillator threshold testing: Measurement of the defibrillation threshold was performed using a modified binary search protocol. This protocol specified three distinct inductions of ventricula
Period: Overall Study
Arm/Group | Pediatric ICD Pts
Started | 20
Completed | 20
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | Pediatric ICD Pts
Number analyzed (Participants) | 20
Age, Continuous [Median (Inter-Quartile Range); unit: years] | 16 [8 to 23]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 7
  Male | 13
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 20
Cardiac diagnosis [Count of Participants; unit: Participants]
  Channelopathy | 11
  Congenital heart disease | 5
  Cardiomyopathy | 4
Weight (kg) [Median (Inter-Quartile Range); unit: kilograms] | 48 [22 to 57]
ICD system configuration [Count of Participants; unit: Participants]
  Transvenous | 12
  Nontransvenous | 8
Location of high-voltage coil [Count of Participants; unit: Participants]
  Transvenous single coil | 7
  Transveous dual coil | 5
  Pericardial | 6
  Subcutaneous | 1
  Pleural | 1
Indication for defibrillation threshold testing [Count of Participants; unit: Participants]
  New implant | 7
  Lead revision | 5
  Generator change | 5
  Surveillance | 3
Anti-arrhythmic medications at testing [Number; unit: participants] — Number of anti-arrhythmic medications and number of subjects did not correlate 1:1, with 5 subjects on >1 anti-arrhythmic agent and some subjects not receiving any anti-arrhythmic agent. For this reason, the total count of anti-arrhythmic medications does not equal the subject number.
  participants
    Beta-blocker | 13
    Calcium-channel blocker | 3
    Amiodarone | 2
    Other | 3

OUTCOME MEASURES:

1. Primary Outcome: Defibrillation Threshold
Description: The defibrillation threshold is a measure of the minimum amount of energy (in Joules) that is able to successfully defibrillate an episode of ventricular fibrillation. This measurement is specific to each individual patient with his/her specific defibrillator configuration. There are several different strategies to measuring this in an individual patient; this study utilized the binary search protocol.
Time Frame: During clinical ICD procedure, as a single event
Measure: Median (Inter-Quartile Range); unit: Joules
Groups:
- Pediatric ICD Pts: Inclusion criteria: 1) weight ≤60 kg, 2) new or existing ICD system, and 3) clinically necessary assessment of the defibrillation efficacy of the ICD system. Transvenous systems utilized a high-voltage ICD coil with active-fixation lead attached to the right ventricular endocardial surface, whereas non-transvenous systems depended upon a high-voltage shocking coil placed within the pericardial, subcutaneous or pleural space. To be included in the post-shock pacing portion of the study, adequate sinus and AV node function had to be present at baseline. Exclusion criteria included 1) tenuous hemodynamic status felt to warrant abbreviation of the defibrillation efficacy testing or 2) inability to induce fibrillation during defibrillation threshold testing (DFT).
Arm/Group | Pediatric ICD Pts
Number analyzed (Participants) | 20
Joules | 7 [4 to 9]

2. Secondary Outcome: Do DFTs Vary by Type of ICD Systems Implanted?
Description: The defibrillation threshold (as measured in Joules as already described in the details regarding the primary outcome) will be compared between patients with two distinct general types of implanted defibrillator systems: 1) transvenous ICD systems (defibrillator leads located inside the vein and attached to the endocardial surface of the heart) and 2) non-transvenous ICD systems (including all other types of debrillation systems).
Time Frame: During clinical ICD procedure, as a single event
Measure: Median (Inter-Quartile Range); unit: Joules
Groups:
- Transvenous ICDs: Patients with an implanted defibrillator system utilizing a transvenous high voltage coil/defibrillator lead.
- Non-transvenous ICDs: Patients with an implanted defibrillator system utilizing a nontransvenous high voltage coil/defibrillator lead.
Arm/Group | Transvenous ICDs | Non-transvenous ICDs
Number analyzed (Participants) | 12 | 8
Joules | 7 [4.5 to 11] | 6 [3.5 to 9]

3. Secondary Outcome: Intrinsic Heart Rate in the Immediate Post-defibrillation Period
Description: A patient will be considered to have an intrinsic slow heart rate in the period of time immediately following defibrillation (20 seconds) if any of the following are observed: >7 paced beats, asystole >4 seconds, or experienced >10% decrease in systolic blood pressure.
Time Frame: During clinical ICD procedure, as a single event
Population: Post-defibrillation episodes in which intrinsic rhythm was evaluable and pacing was necessary
Measure: Number; unit: episodes
Units Other Than Participants: Post-defibrillation episodes
Groups:
- Post-shock Pacing Assessment: In addition to the baseline study inclusion criteria, this arm included only patients who met the additional inclusion criteria of adequate sinus node function and intact AV node conduction.
Arm/Group | Post-shock Pacing Assessment
Number analyzed (Participants) | 16
Number analyzed (Post-defibrillation episodes) | 49
episodes | 0

ADVERSE EVENTS:
Time Frame: Peri-procedural (day of clinincal procedure)
Arm/Group | Pediatric ICD Pts
All-Cause Mortality (participants affected / at risk) | 0/20
Serious Adverse Events (participants affected / at risk) | 0/20
Other Adverse Events (participants affected / at risk) | 0/20

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes